CLINICAL TRIAL: NCT03372564
Title: CREST: A Randomized Controlled Trial Comparing Inter-portal Hip Capsular Repair vs. No Repair Following Hip Arthroscopy
Brief Title: CREST: Capsular Repair During Hip Arthroscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aaron Krych, Professor of Orthopedics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-009462
Record Dates: First submitted 2017-11-27; First posted 2017-12-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hip Arthroscopy
MeSH Terms: interventions — Papaverine; Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Capsule Repair (Experimental): Patients in the intervention group (Hip capsule repair) will undergo initial diagnostic arthroscopy of the hip. Two to three standard portals (anterolateral, mid anterior, distal antero-lateral, posterolateral) will be used during the entire procedure to assess and treat the patient. After establishing standard portals, an interportal capsulotomy is completed to allow for complete evaluation of the central compartment of the hip. In the central compartment, significant and obvious pathologies will be addressed accordingly. Following addressing central compartment pathologies, cam impingement type lesions in the peripheral compartment will be treated. Once all pathologies are addressed, the interportal capsulotomy10 will be repaired by using simple interrupted sutures with absorbable suture (Number 1 Vicryl). Three to four simples sutures will be placed and tied using arthroscopic technique.
  Interventions: Procedure: Hip Capsule Repair
- No Hip Capsule Repair (Control) (No Intervention): Patients in the control group (no hip capsule repair) have the same portals utilized and will have the same interportal capsulotomy performed. They will have all central and peripheral compartment pathologies addressed in the same way that the study group does. At the conclusion of the case, the hip capsule will be left open and not repaired.

INTERVENTIONS:
Procedure: Hip Capsule Repair — In the central compartment, significant and obvious pathologies will be addressed accordingly. Following addressing central compartment pathologies, cam impingement type lesions in the peripheral compartment will be treated. Once all pathologies are addressed, the interportal capsulotomy10 will be repaired by using simple interrupted sutures with absorbable suture (Number 1 Vicryl).
  Arms: Hip Capsule Repair

SUMMARY:
Capsular REpair randomiSed controlled Trial (CREST) is a multi-center, randomized controlled trial with a sample size of 240 patients (120 patients in each group). The primary outcome measure is functional outcome as measured by the change in Hip Outcome Score at 6 months with secondary outcomes being hip range of motion, i-HOT 12, overall satisfaction, and VAS. Patients are stratified based on gender. Patients, outcome assessors, and data analysts are blinded to surgical allocation. Using an intention-to-treat approach, outcome analyses will be performed using an analysis of covariance and descriptive statistics.

DETAILED DESCRIPTION:
Background Femoroacetabular impingement (FAI) is a well-described condition that causes hip pain in young to middle age adults. Cross sectional studies have estimated that the prevalence of hip impingement ranges from 14-17% among asymptomatic young adults and nearly 95% among competitive athletes. FAI occurs as a result of a size and shape mismatch between the femoral head and the acetabulum. There are two subtypes of FAI: Cam type and Pincer type. Cam type is caused by a misshaped femoral head and pincer is caused by an over coverage of the acetabular rim. Most patients have a mixed type of Cam and pincer impingement that involves some degree of an abnormally shaped femoral neck and over coverage of the acetabulum. Arthroscopic treatment for FAI has demonstrated promising results. It has been shown to alleviate pain and improve function with good return to sport rates in young athletes with FAI.

Although arthroscopic treatment for FAI has provided promising results, there is much debate over treatment of the capsule after arthroscopic surgery. Surgeons usually either choose to perform a capsulotomy or a partial capsulectomy during arthroscopic surgery to increase their viewing space in order to perform procedures to address intra-articular pathologies.

The hip capsule is made up of four components: The iliofemoral, pubofemoral, and ischiofemoral ligaments and the zona orbicularis. The iliofemoral has been shown to be the strongest of these ligaments and the most important stabilizer in resisting anterior translation and hip dislocation. During arthroscopic hip surgery, surgeons often use an interportal cut made between the mid-anterior and anterolateral portal to allow visualization of the joint. Surgeons may choose to either leave the capsule open or repair it. As techniques have evolved, more interest has been placed on repairing the capsule in order to improve stability following arthroscopic hip surgery. Frank et al. recently reported that patients undergoing T-capsulotomy with complete closure had improved outcomes compared to patients who received only partial closure. Wylie et al. recently showed improved post-operative patient reported outcomes (PROs) following revision hip arthroscopy in order to repair the capsule.

The goal of the CREST is to evaluate functional stability and patient reported outcome scores following capsular repair after arthroscopic hip surgery for FAI.

Overview of study design

Patients are recruited by experienced hip surgeons for inclusion. Patients will either be randomized to have their capsule repaired upon completion of arthroscopic hip surgery or will have it left unrepaired. Surgeons will measure pre-operative pain and function. Over a 24 month period patients will be evaluated for pain, functional impairment, and activity level.

Patient recruitment and screening The CREST study will be performed at the Mayo Clinic (Rochester, MN and Arizona campus), the American Hip Institute (Chicago, IL). The surgeons coordinating this study have performed over 5,000 hip arthroscopies collectively. They have shown the ability to recruit patients to perform these procedures and demonstrated the ability to follow these patients for 2 years or longer in order to assess outcomes. They are planning to start enrolling patients in January of 2017 and continue the enrollment process on an ongoing basis. Patients will be classified based on three categories: 1) Included in the study and randomized 2) excluded if they do not meet the inclusion criteria, or 3) Missed (patients that were eligible but not included in the study due to an error or limited staff availability at the time of presentation).

Study Follow-Up

Patients will undergo standard of care evaluation at baseline with follow-up at 6 weeks, 3 months, 6 months, 12 months, and 24 months after surgery. Patients who are unable to attend the follow-up appointments will be contact by email via OBERD to complete questionnaires and if this fails they will be contacted by phone.

Minimizing Crossovers

It is very unlikely that there will be crossover between the two groups because both groups will have intra-articular pathology that is causing pain addressed during surgery. Any patient who does crossover, will be analyzed with the group they were randomized (intention to treat analysis).

Protecting against sources of bias

Multiple methods will be implemented to protect against bias. There will be concealment of the randomization, investigators will maximize possible blinding, investigators will utilize strategies to limit loss to follow-up and crossovers, and investigators will objectively adjudicate patient outcomes.

Maximizing Patient Follow-Up

Both sites involved have used OBERD to collect outcomes for the past three years. They have shown the ability to follow patients for many years after surgery using this system. Both sites will have patients complete the PROs on iPads while waiting to be seen before clinical visits to the surgeons. For patients who are unable to come in for clinical visits, OBERD has the capability of sending reminders via email to patients who have not filled their PROs out at the correct follow up time. If both of these strategies fail, then the patients will be contacted on every phone number available in order to achieve maximum follow-up.

Sample size calculation Based on a pilot data previously collected by one of the participating surgeons, investigators used sample size estimation to calculate that 240 total patients (120 patients in each group) would be required to demonstrate a difference in subjective patient reported outcome scores (mHHS and HOS-ADL and HOS-Sports) of the two groups with an effect size of 0.8 with an alpha level of 0.05 and power of 80%. Investigators added a potential 20% loss to follow-up in our calculations, which is very conservative. This would leave 100 patients in each group at final follow-up and 200 patients in the study overall. This was powered to detect a clinically significant difference of 2.0 points in mHHS scoring and 3.84 points in HOS-ADL and HOS-Sports. This is well within previously reported minimal clinically important differences between these three outcome scores.

In addition, investigators will also include equal groups of male and female hips (60 males and 60 females in each group). In this manner, differences between gender will be powered to detect a difference of 4 points for mHHS and 7.72 points for HOS score.

Data Management

Data will be collected in OBERD at both sites. Upon entering data into OBERD, personnel from each site will ensure its accuracy and will discuss and correct all missing, inconsistent, or inaccurate data.

Data Safety and Monitoring Committee

All data will be stored safely at each site and on the OBERD server which has been verified to have the appropriate safe guards for patient privacy. All patients that are exchanged between institutions will have all identifying information removed (name and clinic number) in order to ensure privacy of the patients as well.

Ethics and Institutional Review Board (IRB) Approval

The CREST trial patients will sign an IRB approved consent form that describes this study and provides sufficient information for patients to make an informed and educated decision about their participation in the study. All participating institutions will obtain IRB approval from the institution for study protocol, the consent form template, the PROs, and any additional protocol items. Any amendments to the protocol will be communicated to the head site (Mayo Clinic) primary investigator (Dr. Aaron Krych).

All study and patient information will be kept private and only be accessed by staff involved in the study. All paper charts will be kept in secure, locked cabinets and all electronically stored documents will be stored on secure databases that have received approval from both institutions software security advisors. Information exchanged between sites involving patient information will have all identifiers removed to preserve privacy.

Discussion

The CREST trial is necessary because as hip arthroscopy continues to grow in popularity as the primary treatment for FAI there will be continued debate on how to handle the hip capsule after surgery, unless studies like this are performed. There is still no compelling evidence on the importance of hip capsule repair following arthroscopic hip surgery. Randomized controlled trials like the CREST trial are the only feasible way to determine its importance and determine if there is a difference in clinical outcomes following hip arthroscopy in patients who receive a capsular repair versus those who do not.

The CREST trial is the first RCT to evaluate the difference in outcome in patients who receive capsular repair versus those who do not following hip arthroscopy. This trial will help overcome many of the biases that currently drive the literature and current evidence for capsular repair. The study will be designed to have significant power to determine a clinically important difference between the two groups in regards to clinical and functional outcomes. The surgeons involved in the study have already shown the ability to recruit patients to trials and the ability to follow these patients, having a collective 5,000 patients with outcomes stored in a shared database already.

This trial, like all surgical RCTs, have some limitations that cannot be avoided. First, although all surgeons are fellowship trained and considered to be experts in hip arthroscopy and the treatment in FAI, there are differences in surgical techniques and intra-operative decision making that cannot be normalized. However, this also makes the results of this RCT more generalizable. Also, as with any RCT, the surgeons cannot be blinded to the treatment allocation.

The vast increase in surgical treatment of FAI has mainly consisted of retrospective studies assessing its efficacy. Even fewer studies have looked at hip capsular repair and its role following hip arthroscopy for FAI. The CREST trial will be the first randomized controlled trial to assess clinical and functional outcome differences in patients who have their hip capsule repaired versus unrepaired following hip arthroscopy for symptomatic hip pathology.

ELIGIBILITY:
Criteria: Inclusion Criteria:

1. Adults aged 18 to 50 (men or women)
2. Hip pain for greater than 3 months that has failed non-operative treatment (physical therapy, NSAIDS, rest)
3. FAI documented on X-Ray or Magnetic resonance imaging (MRI) or magnetic resonance arthrogram (MRA)
4. Intraoperative labral repair or intact labrum
5. Informed consent from the participant
6. Ability to comprehend and speak English and the study design.

Pre-operative exclusion criteria are the following:

1. Hypermobility/Ehlers-Danlos syndrome
2. Evidence of hip dysplasia (Center edge angle less than 20)
3. Previous surgery or trauma of the affected hip
4. Severe acetabular deformities such as circumferential labral ossification, acetabular protrusion20
5. Inflammatory/ autoimmune disease
6. Immunosuppressant medication
7. Significant medical co-morbidities such as uncontrolled diabetes, hypertension, congestive heart failure, etc.
8. Severe mental or physical disability requiring assistance in daily living
9. History of pediatric hip disease with previous operation (developmental dysplasia, Legg-Calve-Perthes, Slipped capital femoral epiphysis)
10. Presence of advanced hip osteoarthritis (Tonnis grade 2 or 3)18
11. Worker's compensation status
12. Intraoperative microfracture, or other procedure that would alter postoperative rehabilitation
13. Intraoperative labral debridement or labral reconstruction
14. Peri-trochanteric or deep gluteal space arthroscopy
15. Avascular necrosis

Intra-operative exclusion criteria are the following:

1. Labral debridement
2. Labral reconstruction
3. Poor quality capsular tissue
4. Hyperlaxity based on excessive subluxation of the joint greater than 2 cm with standard 50 pounds of traction
5. Concomitant procedures such as MFX and iliopsoas lengthening will be included

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-11-07 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Hip Function | Baseline, 6 months
  The main outcome assessed will be hip function including change in percentage of Hip outcome score (HOS score) from baseline to 6 month follow-up. The subscale of ADL (activities of daily living) and Sport will be utilized. each HOS subscale is calculated from 0 to 100%, with 100% being the best score.

SECONDARY OUTCOMES:
Hip ROM | Baseline, 6 months
  Hip range of motion will be assessed by a blinded examiner. The change in degrees of range of motion from baseline to 6 month examination will be assessed.
Visual Analog Pain Score Progression | Baseline, 6 months
  The change in pain scores will be assessed using VAS (visual analog scale) pain score, analyzing the change in units of measure between the baseline and 6 month time-points.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Krych, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - American Hip Institute, Westmont, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domb BG, Stake CE, Finley ZJ, Chen T, Giordano BD. Influence of capsular repair versus unrepaired capsulotomy on 2-year clinical outcomes after arthroscopic hip preservation surgery. Arthroscopy. 2015 Apr;31(4):643-50. doi: 10.1016/j.arthro.2014.10.014. Epub 2014 Dec 16. PMID 25530511
- [Background] Frank RM, Lee S, Bush-Joseph CA, Kelly BT, Salata MJ, Nho SJ. Improved outcomes after hip arthroscopic surgery in patients undergoing T-capsulotomy with complete repair versus partial repair for femoroacetabular impingement: a comparative matched-pair analysis. Am J Sports Med. 2014 Nov;42(11):2634-42. doi: 10.1177/0363546514548017. Epub 2014 Sep 11. PMID 25214529
- [Result] Wylie JD, Beckmann JT, Maak TG, Aoki SK. Arthroscopic Capsular Repair for Symptomatic Hip Instability After Previous Hip Arthroscopic Surgery. Am J Sports Med. 2016 Jan;44(1):39-45. doi: 10.1177/0363546515608162. Epub 2015 Sep 29. PMID 26419897
- [Result] Chahal J, Van Thiel GS, Mather RC 3rd, Lee S, Song SH, Davis AM, Salata M, Nho SJ. The Patient Acceptable Symptomatic State for the Modified Harris Hip Score and Hip Outcome Score Among Patients Undergoing Surgical Treatment for Femoroacetabular Impingement. Am J Sports Med. 2015 Aug;43(8):1844-9. doi: 10.1177/0363546515587739. Epub 2015 Jun 15. PMID 26078452
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials